CLINICAL TRIAL: NCT05887531
Title: Effectiveness of a Prehabilitation Consultation in Self-care and Physical Exercise in Patients Diagnosed With Abdominopelvic Cancer
Brief Title: Abdominopelvic Cancer Prehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Principal Investigator, María Pilar Suárez Alcázar, Principal Investigator, Universitat Jaume I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: malcazar
Record Dates: First submitted 2023-05-15; First posted 2023-06-02 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Prehabilitation; Cancer of Colon; Cancer of Rectum; Cancer, Ovarian
Keywords: Selfcare; Fisical exercice; Prehabilitation
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Ovarian Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation (Experimental)
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — Patients will be included in a prehabilitation program

SUMMARY:
The main objective of this research is to determine the effectiveness of a Prehabilitation consultation in self-care and physical exercise aimed at patients diagnosed with abdominopelvic cancer with initial surgical indication as part of their therapeutic plan.

ELIGIBILITY:
Inclusion Criteria:

* Majority (greater than or equal to 18 years).
* Diagnosis of abdominopelvic cancer and initial surgical indication as part of its therapeutic plan from the General Surgery Services of the General University Hospital of Castellón.
* Ability to give informed consent.

Exclusion Criteria:

* Inability to understand the information provided or insufficient knowledge of the Spanish language.
* Inability to carry out the scheduled intervention according to the physician's criteria.
* Neoadjuvant treatment to colorectal surgery.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Post-surgical recovery time | More than 2 days
  To determine if there is a reduction in post-surgical recovery time until the start of adjuvant therapy in patients with abdominopelivoc cancer after their incorporation into the Prehabilitation program in self-care and directed physical exercise.
Post-surgical readmisions | until 4 weeks from surgery
  To determine if there is a reduction in the number of readmisions in patients with abdominopelvic cancer after their incorporation into the Prehabilitation program in self-care and directed physical exercise.

SECONDARY OUTCOMES:
Self-care capacity | before surgery
  To know if there is an improvement in the self-care capacity mesured by the Appraisal of Self-care Agency Scale (ASA) scale in patients with abdominopelvic cancer after their incorporation into the Pre-habilitation program in self-care and directed physical exercise. Minimum value: 24 y Maximum value: 96. Higher scores mean a better outcomes.
Anxiety levels | before surgery
  To establish whether there is a decrease in preoperative anxiety levels mesured by Hospital Anxiety and Depression Scale in patients with abdominopelvic cancer after their incorporation into the Prehabilitation program in self-care and directed physical exercise.
Aerobic capacity | before surgery
  To determine if there is an improvement in aerobic capacity mesured by walking test in patients with abdominopelvic cancer after their incorporation into the Prehabilitation program in self-care and directed physical exercise. Higher scores mean a better outcomes.
Flexibility | before surgery
  To determine if there is an improvement flexibility mesured by set and reach test in patients with abdominopelvic cancer after their incorporation into the Prehabilitation program in self-care and directed physical exercise. Higher scores mean a better outcomes.
Strength | before surgery
  To determine if there is an improvement strength mesured by hand grip in patients with abdominopelvic cancer after their incorporation into the Prehabilitation program in self-care and directed physical exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Suárez María Pilar, Principal Investigator — Universitat Jaume I
Locations (1):
- Universitat Jaume I, Castellon, Castellón, Spain